CLINICAL TRIAL: NCT00089063
Title: A Randomized Phase II Continuation Booster Trial After A Vaccine Combining Tyrosinase/GP100/Mart-1 Peptides Emulsified With Montanide ISA 51 and ISA 51 VG With Or Without GM-CSF For Patients With Resected Stages IIB/C, III And IV Melanoma
Brief Title: Vaccine Therapy With or Without Sargramostim in Treating Patients Who Have Undergone Surgery for Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02618; NCI-2012-02618 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LAC-USC-042011; NCI-6618; LAC-USC-0A1033; CDR0000378033; 10M-03-8 (Other: University of Southern California); 6618 (Other: CTEP)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2013-10

CONDITIONS: Ciliary Body and Choroid Melanoma, Medium/Large Size; Extraocular Extension Melanoma; Iris Melanoma; Stage IIB Melanoma; Stage IIC Melanoma; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — MART-1 Antigen; incomplete Freund's adjuvant; montanide ISA 51; sargramostim

ARMS (2):
- Arm I (vaccine therapy) (Experimental): Patients receive vaccination comprising tyrosinase peptide, gp100 antigen, and MART-1 antigen emulsified with Montanide ISA-51 and ISA-51 VG SC on day 1 of weeks 0, 26, 52, 78, and 104 (total of 5 vaccinations).
  Interventions: Biological: tyrosinase peptide; Biological: gp100 antigen; Biological: MART-1 antigen; Biological: incomplete Freund's adjuvant; Drug: Montanide ISA 51 VG; Other: laboratory biomarker analysis
- Arm II (vaccine therapy, sargramostim) (Experimental): Patients receive vaccination comprising tyrosinase peptide, gp100 antigen, and MART-1 antigen emulsified with Montanide ISA-51 and ISA-51 VG as in arm I. Patients also receive sargramostim (GM-CSF) SC on days 1-5 of weeks 0, 26, 52, 78, and 104.
  Interventions: Biological: tyrosinase peptide; Biological: gp100 antigen; Biological: MART-1 antigen; Biological: incomplete Freund's adjuvant; Drug: Montanide ISA 51 VG; Biological: sargramostim; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: tyrosinase peptide — Given SC
Biological: gp100 antigen — Given SC
Biological: MART-1 antigen — Given SC
Biological: incomplete Freund's adjuvant — Given SC
Drug: Montanide ISA 51 VG — Given SC
Biological: sargramostim — Given SC
  Arms: Arm II (vaccine therapy, sargramostim)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying vaccine therapy and sargramostim to see how well they work compared to vaccine therapy alone in treating patients who have undergone surgery for stage IIB, stage IIC, stage III, or stage IV melanoma. Vaccines made from peptides may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim increase the number of immune cells found in bone marrow or peripheral blood. Combining vaccine therapy with sargramostim may make a stronger immune response.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate immune reactivity to a tyrosinase:368-376 (370D) /gp100: 209-217 (210M)/MART-1 26-35 (27L) peptide vaccine with Montanide ISA 51 with or without GM-CSF administered as a booster for five vaccinations over two years.

OUTLINE: This is a randomized, parallel, continuation study. Patients are stratified according to response to prior vaccination (response to 1 peptide vs response to 2 or more peptides). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive vaccination comprising tyrosinase peptide, gp100 antigen, and MART-1 antigen emulsified with Montanide ISA-51 and ISA-51 VG subcutaneously (SC) on day 1 of weeks 0, 26, 52, 78, and 104 (total of 5 vaccinations).

Arm II: Patients receive vaccination comprising tyrosinase peptide, gp100 antigen, and MART-1 antigen emulsified with Montanide ISA-51 and ISA-51 VG as in arm I. Patients also receive sargramostim (GM-CSF) SC on days 1-5 of weeks 0, 26, 52, 78, and 104.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed at 2-4 weeks, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients (20 per treatment arm) will be accrued for this study within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed protocol 10M-01-1 or 10M-00-4 are eligible for this study provided that

  * They have received all injections with evidence of an immune response
  * They have not experienced recurrence of the melanoma
  * Not more than twelve months have elapsed since the final injection on either protocol
  * They experienced no grade 3 or 4 toxicity attributed to the prior vaccine regimen
* Serum creatinine of 2.0 mg/dl or less
* Total bilirubin of 2.0 mg/dl or less
* SGOT/SGPT of 2.5 X institutional norm or less
* Total WBC of 3,000 or more
* At least 1500 granulocytes
* Hemoglobin of 9.0 gm/dl or more
* Platelet count of 100,000 per cu mm. or more
* ECOG performance status of 0 or 1
* Patients will be eligible for this trial if they have failed alpha-interferon, if it is felt to be contraindicated due to a pre-existing medical or psychiatric condition or if they have refused treatment with it
* Ability to read, understand and willingness to sign an IRB-approved informed consent
* Patients who have had another malignancy but with no evidence of disease for greater than 5 years from accrual to the current trial will be eligible if it is felt they are likely to be cured; patients with squamous or basal carcinoma of the skin or carcinoma in situ of the cervix that have been treated with curative intent can be accrued to this trial 30 days after treatment

Exclusion Criteria:

* Who have undergone any other systemic therapy for their melanoma, including radiation therapy since completion of 10M-01-1 or 10M-00-4
* Have major systemic infections like pneumonia or sepsis, coagulation or bleeding disorders, or other major medical illnesses of the gastrointestinal, cardiovascular or respiratory systems
* Who require systemic, ocular or inhaled corticosteroids
* Who are pregnant or lactating, since the risk of autoimmune reactivity to tyrosinase, MART-1 or gp100 is felt to present a risk to the fetus or a breast feeding infant; effective birth control for men and women is required during and for four months after the study is finished
* Who are known to be positive for hepatitis BsAg, hepatitis C antibody or HIV antibody; since cells removed for ex vivo handling and tissue culture cannot be virus positive, and the effects of melanoma peptides might be detrimental to HIV positive patients, patients positive for the above viruses will not be treated on this trial
* Who have had a known allergic reaction to GM-CSF, Montanide ISA 51 (IFA) or any of the peptides included in this protocol
* Who have a prior history of uveitis or autoimmune inflammatory eye disease, immune hemolytic anemia or other active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Immune response | Baseline
  Summarized using means and confidence intervals (after transformation to render the data compatible with the assumptions of the normal distribution).
Immune response | Week 106
  Summarized using means and confidence intervals (after transformation to render the data compatible with the assumptions of the normal distribution).

SECONDARY OUTCOMES:
Disease-free survival | Up to 2 years
  Kaplan-Meier curves will be drawn to display the survival and time to recurrence. The log-rank test and estimates of relative risk based on the log-rank statistics will be performed. 95% confidence intervals will be constructed for the median DFS and OS.
Overall survival | Up to 2 years
  Kaplan-Meier curves will be drawn to display the survival and time to recurrence. The log-rank test and estimates of relative risk based on the log-rank statistics will be performed. 95% confidence intervals will be constructed for the median DFS and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weber, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States